CLINICAL TRIAL: NCT06909227
Title: Relevance of Veinous Lactates Dosage at the End of a Surgical Procedure to Predict Postoperative Complications in Children 0-1 Years
Brief Title: Relevance of Veinous Lactates to Predict Postoperative Complications in Children 0-1 Years
Acronym: PLANN
Status: Recruiting | Type: Observational
Sponsor: Hôpital Armand Trousseau (Other)
Responsible Party: Principal Investigator, Pr Isabelle CONSTANT, Professor of Anesthesiology, Head of Department, Hôpital Armand Trousseau
Other Study IDs: PLANN
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: General Anesthesia; Infant
Keywords: pediatric; anesthesia; lactate; complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- infants 0-1 years undergoing surgery under general anesthesia: Not including day-case surgery, or cardiac surgery
  Interventions: Procedure: surgery under general anesthesia

INTERVENTIONS:
Procedure: surgery under general anesthesia — Only in children, < 1 year old non-cardiac surgery

SUMMARY:
This study will investigate if the dosage of veinous lactate at the end of a surgical procedure is related to post-operative complications occurring within 3 months in young infants aged 0-1 years.

Blood samples are acquired routinely before emergence of general anesthesia, from the IV line put in place for anesthesia.

The investigators hypothesized that elevated lactates would be associated with more postoperative complications in this population, as is the case in adults.

ELIGIBILITY:
Inclusion Criteria:

* surgery under general anesthesia
* age < 1 year

Exclusion Criteria:

* ambulatory surgery
* cardiac surgery
* preoperative hemodynamic instability
* Weight < 2 kg

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children requiring a surgical procedure
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Post-operative complications occurring within 3 months after surgery | within 3 months after surgery
  ICU admission Re-operation Re-admission Death

CONTACTS AND LOCATIONS:
Overall Officials: Nada Sabourdin, MD, PhD, Study Director — Armand Trousseau University Hospital; Isabelle Constant, MD, PhD, Study Chair — Armand Trousseau University Hospital
Locations (1):
- Armand Trousseau University Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided
Will have to check adherence to confidentiality protocols.

REFERENCES:
- [Background] Zheng D, Yu GL, Zhou YP, Zhang QM, Wang CG, Zhang S. Association between lactic acidosis and multiple organ dysfunction syndrome after cardiopulmonary bypass. PeerJ. 2024 Jan 31;12:e16769. doi: 10.7717/peerj.16769. eCollection 2024. PMID 38313014
- [Background] Stephens EH, Epting CL, Backer CL, Wald EL. Hyperlactatemia: An Update on Postoperative Lactate. World J Pediatr Congenit Heart Surg. 2020 May;11(3):316-324. doi: 10.1177/2150135120903977. PMID 32294015